CLINICAL TRIAL: NCT01899820
Title: Evaluation of the Efficacy of Artemisinin Combination Therapy in Kenya
Acronym: EAPHLNP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sabah Ahmed Omar (Other)
Collaborators: World Bank (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Sabah Ahmed Omar, Centre Director of KEMRI CGMR-C and Study Principal Investigator, KEMRI-Wellcome Trust Collaborative Research Program
Organization: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEMRI_CT_2013/0017; SSC 2276 (Other: KEMRI Scientific Steering Committee)
Record Dates: First submitted 2013-04-17; First posted 2013-07-15 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemether lumefantrine (Active Comparator): Tablets, 1-4 tablets (weight calculated dose), BD, at hr 0, 8, 24, 36, 48 and 60.
  Interventions: Drug: Artemether lumefantrine
- Dihydroartemisinin piperaquine (Experimental): Tablets, 2 paediatric tablets/1 adult tablet, OD, every 24 hours for 48 hours
  Interventions: Drug: Dihydroartemisinin piperaquine

INTERVENTIONS:
Drug: Artemether lumefantrine — Artemether 20mg Lumefantrine 120mg
  Other Names: Coartem
  Arms: Artemether lumefantrine
Drug: Dihydroartemisinin piperaquine — Dihydroartemisinin 20mg Piperaquine 160mg
  Other Names: Duocortexin
  Arms: Dihydroartemisinin piperaquine

SUMMARY:
Artemisinin-based combination therapies (ACTs) are recommended for use against uncomplicated malaria in areas of multi-drug resistant malaria. The Ministry of Health, Division of Malaria Control (DOMC) rolled out the use of artemether-lumefantrine as the first line treatment for uncomplicated malaria in 2006.The development of the ACTs and its derivatives are the most rapidly acting of all the current antimalarial drugs and recognition of their potential role as a component of combination therapy have led to several large trials aimed at assessing different combinations of existing drugs, and to the specific development of new combination drugs.

This proposal aims to (1) evaluate the efficacy of artemisinin-based anti-malaria combination drugs in different sites across Kenya (2) elucidate the markers of resistance to ACTs through molecular genetics and in this process further strengthen capacity in the proposed study sites as well as improve links between research and control ultimately to influence malaria treatment policy and practice.

Five groups in East Africa will conduct a multi-centre, randomised, two arm trial to assess the efficacy of dihydroartemisin-piperaquine with artemether-lumefantrine as the comparative drug. The network will determine antimalarial drug efficacy using standardised protocols and collate clinical responses and adverse events. Molecular markers to artemisinin resistance will be investigated by molecular sequencing and comparison of parasite profiles in drug failure cases. Recrudescence or re-infections will be differentiated by analysis of the MSP1, MSP2 and GLURP genes and assess transmission dynamics post treatment. Data from these studies will be captured into a database developed by the network. The latter offers several advantages including

* Working towards the standardization of methodologies and common protocols as a way of comparing data across sites
* Pulling together datasets and conduct a multi-centre analysis
* Sharing and coordinating quality assurance mechanisms

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 months - 5 years (in high endemic areas); 6 months to 10 years (in low endemic areas) inclusive.
2. Presence of axillary temperature > 37.5oC or rectal / tympanic temp > 38.0oC, or history of fever in the last 24 hours.
3. Monoinfection with Plasmodium falciparum with parasitaemia, asexual parasitemia between 2,000 - 200,000 p/µl (in areas of high transmission); 1,000-100,000p/ µl (in areas of low to moderate malaria transmission)
4. Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
5. Signed informed consent form by the parents or legal guardian.

Exclusion Criteria:

1. Presence of clinical danger signs: not able to drink or breast-feed, vomiting (>twice in 24 hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand;
2. Mixed or mono-infection with another Plasmodium species detected by microscopy;
3. Presence of co-morbid infection (e.g. acute lower respiratory tract infection, severe diarrhoea with dehydration, Severe Anaemia) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases,Epilepsy, HIV/AIDS);
4. History of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s).

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the PCR-corrected and parasitological response (PCR corrected ACPR) at days 28 and 42. Change in this outcome measure will be assessed. | Day 28 and day 42
  ACPR is defined as the absence of parasitaemia on day 42 irrespective of the temperature without previously meeting any of the criteria of early treatment failure or late clinical or parasitological failure.
  Patients with late asexual parasite reappearance will be considered ACPR if the CR analyses shows a new infection rather than a recrudescence (through PCR genotyping).
  The total treatment failure is defined according to the WHO criteria as the sum of early and late treatment failures.

SECONDARY OUTCOMES:
Crude (PCR uncorrected) ACPR ratio at day 28 (PCR uncorrected ACPR) | Day 28
Cure ratios at day 28, 42, (PCR corrected and PCR uncorrected). Change in this outcome measure will be assessed. | Day 28 and day 42
Fever Clearance Time (FCT) | 0 to 48 hours
  This will be defined as the time (hrs) from the start of a patient's treatment to the first consecutive axillary temp measurements below 37.5 for at least 48 hrs
Asexual parasite clearance time (PCT) | Day 0 to day 28, upto day 42
  PCT(proportion of patients remaining parasitaemic) defined as the time (in hours) from the start of a patient's treatment to 2 consecutive negative blood slides (collected at different days)
Gametocyte carrier rates and geometric mean densities (excluding negatives) will be compared on days 7, 14, 28 and 42. Change in this outcome measure will be assessed. | Day 7, 14, 28 and 42
Changes of haemoglobin (Hb) concentration from day 0 to days 28, and 42 | Day 0, day 28 and day 42
Number of participants with adverse events | Up to day 42
Comparison between adverse events related to artemether lumefantrine and dihydroartemisinin piperaquine | Up to day 42
Temperature | Up to day 42
Oxygen saturation | Up to day 42
Heart rate | Up to day 42
Respiratory rate | Up to day 42

CONTACTS AND LOCATIONS:
Overall Officials: Sabah A Omar, PhD, Principal Investigator — KEMRI CGMR-C
Locations (7):
- Kenya (7):
  - Busia district hospitals, Busia, Busia County
  - Kisii district hospitals, Kisii, Kisii County
  - Kitale district hospitals, Kitale, Kitale
  - Msambweni sub-district hospital, Msambweni, Kwale County
  - Machakos district hospital, Machakos, Machakos County
  - Malindi district hospitals, Malindi, Malindi
  - Nyando district hospital, Nyando, Nyando